CLINICAL TRIAL: NCT05866549
Title: The Effect of The Mindfulness-based Childbirth and Parenting Program on Prenatal Attachment and Depression, Stress, Anxiety Levels of Pregnants
Brief Title: The Effect of The Mindfulness-based Childbirth and Parenting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ezgi Findik (Other)
Responsible Party: Sponsor-Investigator, Ezgi Findik, Dr, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20/198
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Mindfulness-based Childbirth and Parenting Program
- Control Group (No Intervention)

INTERVENTIONS:
Other: Mindfulness-based Childbirth and Parenting Program — Mindfulness-based childbirth and parenting program will be applied to individuals in this group. The program consists of nine sessions, eight of which will take place during pregnancy. Sessions planned during pregnancy will be held once a week, lasting 8 weeks.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to determine the effect of Mindfulness-based childbirth and parenting program on prenatal attachment and depression, stress and anxiety levels of pregnants.

The study will be carried out in two different groups. After the pregnants are evaluated in terms of eligibility criteria for the research, the pregnants who are eligible will be informed about the research and written informed consent will be obtained from the pregnants who accept. The random distribution of pregnants to the study groups will be carried out random. The following applications will be made to the groups.

ELIGIBILITY:
Inclusion Criteria:

* Being at 20-30 weeks of gestation
* Being nulliparous

Exclusion Criteria:

* History of psychiatric illness
* Follow-up in the risky pregnancy clinic
* Not completing the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Prenatal Attachment Inventory | immediately after participants are assigned to groups and eight weeks later
  The scale, which is a four-point Likert-type scale, consists of 21 items. A minimum of 21 and a maximum of 84 points can be obtained from the scale. The change in the score obtained by the pregnant indicates that the level of attachment also increases.
Depression Anxiety Stress Scale- 21 (DASS 21) | immediately after participants are assigned to groups and eight weeks later
  In this scale (DASS-21), there are 7 questions each to measure the dimensions of depression, stress and anxiety. The scale is a 4-point Likert Type Scale; 0 -3. Depression, anxiety and stress scores are measured by summing the scores of the related items. A minimum of 0 and a maximum of 21 points can be obtained in each dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Cebeci Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Findik E, Yilmaz Sezer N, Aker MN, Badur D. The effects of the Mindfulness-Based Childbirth and Parenting Program (MBCP) on prenatal attachment, depression, stress, and anxiety in pregnant women: A randomized controlled trial. J Affect Disord. 2025 May 1;376:341-346. doi: 10.1016/j.jad.2025.02.030. Epub 2025 Feb 15. PMID 39961443